CLINICAL TRIAL: NCT02893527
Title: Implementation and Evaluation of a Social Journey Accompanied for Women With Breast Cancer Diagnosis
Brief Title: Implementation and Evaluation of a Social Journey Accompanied in Breast Cancer Diagnosis (EPARS SEIN)
Acronym: EPARS-SEIN
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: An IDMC validated the premature termination of the study on 19/02/2016 for lack of inclusion, with continuation of the FU initially planned for women included
Sponsor: Institut du Cancer de Montpellier - Val d'Aurelle (Other)
Collaborators: Cemka-Eval (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: ICM-URC-2014/33
Record Dates: First submitted 2016-08-29; First posted 2016-09-08 (Estimated); Last update posted 2020-08-10 (Actual); Status verified 2020-08

CONDITIONS: Breast Cancer
MeSH Terms: conditions — Breast Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Group "intervention" (Experimental): Personalized coaching coordinated by a coordinating nurse on a shutdown period of 8 months (consecutive stops).
  Interventions: Behavioral: personalized coaching
- Group "standard" (No Intervention): conventional support

INTERVENTIONS:
Behavioral: personalized coaching — personalized coaching coordinated by a coordinating nurse on a shutdown period of 8 months (consecutive stops).
  Arms: Group "intervention"

SUMMARY:
Evaluate and compare the return to work rate at 12 months

DETAILED DESCRIPTION:
Evaluate and compare the return to work rate at 12 months (from J1C1 [first day of the first adjuvant chemotherapy regimen]) between the "intervention" group (which has accompanied the career) and the standard group course

ELIGIBILITY:
Inclusion Criteria:

* Patient major> 18
* Have a diagnosis of localized breast cancer requiring surgery immediately adjuvant therapy sequence including chemotherapy and radiotherapy
* Being more than 3 years of retirement at diagnosis
* Have a work contract valid at the time of diagnosis (before surgery)
* Do not practice a profession
* Be in possession of his rights (excluding guardianship, curatorship)
* Raise the general social security scheme and have rights to cash benefits in the Languedoc-Roussillon region

Exclusion Criteria:

* Patient minor
* Patient diagnosed with metastatic breast cancer
* Patients refusing to sign the consent
* Patients do not have sufficient understanding of the French language
* Patients for whom it is impossible to give clear information

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 11 (Actual)
Dates: Start 2015-02-24 (Actual); Primary Completion 2016-12 (Actual); Study Completion 2017-12 (Actual)

PRIMARY OUTCOMES:
Evaluate and compare the return to work rate | through study completion, an average of 5 years
  Evaluate and compare the return to work rate at 12 months (from J1C1 [first day of the first adjuvant chemotherapy regimen]) between the "intervention" group (which has accompanied the career) and the standard group course

SECONDARY OUTCOMES:
describe the conditions of the resumption of work | through study completion, an average of 5 years
  The study will also allow to describe the conditions of the resumption of work in 12 months for the patients concerned and to compare these conditions between the 2 groups

CONTACTS AND LOCATIONS:
Overall Officials: William JACOT, Study Chair — Institut régional du Cancer de Montpellier
Locations (1):
- Institut réginal du Cancer de Montpellier, Montpellier, France

IPD SHARING:
Plan to Share IPD: No